CLINICAL TRIAL: NCT04048265
Title: Study of rTMS in the Treatment of Early/Moderate Parkinson's Disease With Pain.
Brief Title: TMS Treatment in Parkinson's Disease With Pain.
Acronym: TMSPDP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Piu Chan, Director, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: chen biao
Record Dates: First submitted 2019-08-06; First posted 2019-08-07 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2019-05

CONDITIONS: Transcranial Magnetic Stimulation; Parkinson Disease; Pain
Keywords: TMS; Parkinson's disease; pain
MeSH Terms: conditions — Parkinson Disease; Pain | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pain in PD Arm one (Experimental): This arm will receive a total 5 sessions of TMS stimulation in a week. Pre and post intervention scales will be performed on week one, week 2 and week 4.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Pain in PD Arm two (Sham Comparator): This arm will receive a total 5 sessions of sham-TMS stimulation in a week. Pre and post intervention scales will be performed on week one, week 2 and week 4.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Transcranial magnetic stimulation (TMS) is a non-invasive method that uses electromagnetic induction to produce electric currents in the cortex that are strong enough to depolarise neurons sufficiently to trigger action potentials. It is an outpatient based procedure that when used in conjunction with a neuro-navigation system, specific cortical areas can be targeted for greater accuracy and efficacy. In clinical studies, TMS is delivered as trains of pulses (repetitive TMS, rTMS) to prolong its effects. While the exact mechanism of TMS-induced analgesia is unknown, it is thought to regulate the activity of the complex cortical and subcortical networks involved in the processing of painful signals and possibly strengthening the endogenous descending pain modulation system

SUMMARY:
Transcranial magnetic stimulation (TMS) is a procedure that has been shown to improve pain in chronic sufferers. It is a well-tolerated procedure that can be performed on an outpatient basis. It uses a plastic covered coil that sends a magnetic pulse through the skull into the brain and by targeting particular areas in the brain it can be used to help modulate the perception of pain.

The study intends to use this technique to treat such a disabling symptom in patients who suffer from Parkinson's Disease (PD). Initially the aim is to study this technique in 48 patients who are suffering from pain and have PD. These patients would require an EEG before and after the stimulation. The stimulation would be performed over ten sessions and the patients would be assessed by a clinician using well recognized clinical tools.

It is anticipated that there will be a meaningful improvement in pain. It is also anticipated that TMS is a safe technique to use in patients with PD. The study will be used to help plan a future study that compares TMS with sham technique to prove whether TMS could be an option in the treatment of such a disabling condition.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Parkinson's disease diagnosed as "clinically confirmed" or "very likely" according to the 2015 MDS clinical diagnostic criteria;
2. Age ≥ 18 Aged ≤ 80 years old;
3. PD patients with pain, exclude tumors, diabetes, osteoarthritis, rheumatoid rheumatism and other diseases, the use of analgesic drugs is not effective or insignificant.
4. After treatment with anti-Parkinson's disease drug regimen, anti-anxiety and depression, sleep drugs, analgesic drugs, etc. for ≥ 14 days, and the dosage is maintained during the treatment;
5. Ability to follow research plans and visit plans.

Exclusion Criteria:

1. Secondary Parkinson's syndrome caused by vascular factors, toxins, drugs, etc., or Parkinson's superposition syndrome.
2. PD patients with persistent head tremors.
3. Dementia, simple intelligent state check (mmse) ≤ 24 points.
4. Patients with suicidal tendencies and psychotic symptoms. 5, previously accepted dbs or damage surgery.

6. Contraindications for TMS (such as history of seizures, pregnant women, installation of pacemakers, metal inclusions in the body, intracranial hypertension, severe bleeding tendency, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Changes in the pain caused by Parkinson's Disease as measured by Visual Analogue Scale Score. | Pre-treatment, post-treatment 0, 4 weeks
  To quantify changes of the severity of pain.

SECONDARY OUTCOMES:
Changes in the patient's parkinson's disease as measured by Unified Parkinson's Disease Rating Scale III(UPDRS III) score. | Pre-treatment, post-treatment 0, 4 weeks
  To quantify changes of the severity of the motor symptoms of Parkinson's Disease.

CONTACTS AND LOCATIONS:
Overall Officials: Biao Chen, MD,PHD, Study Chair — Xuanwu Hospital of Capital Medical University
Locations (1):
- The Neurology Department of Xuanwu Hospital,Capital Medical University, Beijing, Beijing Municipality, China